CLINICAL TRIAL: NCT05897177
Title: Investigating the Pathophysiological Nature of Homosexuality Patients in Egypt, England, China, and Mexico: Multicenter Study.
Brief Title: Investigating the Pathophysiological Nature of Homosexuality
Status: Not yet recruiting | Type: Observational
Sponsor: Mostafa Bahaa (Other)
Collaborators: Mostafa Mahmoud Bahaa Clinical Pharmacy Department, Horus University, New Damietta, Egypt (Unknown)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Teaching assisstant, Tanta University
Organization: Tanta University (Other)
Other Study IDs: 3255
Record Dates: First submitted 2023-05-28; First posted 2023-06-09 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal patients
  Interventions: Behavioral: Subjective Scale of Stigma and Discrimination (SISD).
- Observational group
  Interventions: Behavioral: Subjective Scale of Stigma and Discrimination (SISD).

INTERVENTIONS:
Behavioral: Subjective Scale of Stigma and Discrimination (SISD). — Subjective Scale of Stigma and Discrimination (SISD) A sixdimension self-administered scale will be used that included statements with which the participants agreed or disagreed. The scale consists of 23 Likert-type items and responses range from 1 ("completely in disagreement") to 5 ("completely in agreement"), grouped together to represent the six indicators making up this part of the scale

SUMMARY:
Debate continues on whether or not male homosexuality (MH) is a result of biological or cultural factors. The debate persists despite the fact that these two sides have different abilities to create a scientific environment to support their cause. Biological theorists produced evidence, however, that these are not always robust. On the other hand, social theorists, without direct evidence confirming their positions, criticize, with good argument, methods and results of the other side.

DETAILED DESCRIPTION:
Is there anything more controversial than homosexuality and its origin? Despite the evidence that bisexual or homosexual behaviour is largely practiced in nature, in close to 1,500 species no less, ranging from primates to gut worms [4], the majority of religious authorities, as well as some political institutions, consider sex with people of the same gender unnatural. Confusion between the level of biological evidence with the level of moral and metaphysic aspects has been and is, unfortunately, frequent. However, we can immediately answer the question in the title: yes, definitively, homosexuality is natural. Would this suggest that biology plays a major role in homosexuality? Probably, but not necessarily. While some people believe that sexual orientation is innate and fixed, for others, sexual orientation may develop across a person's lifetime. The words of John Bancroft, which conclude this Controversy, clarify several aspects of these opposite interpretations 5.

Controversy is limited to male homosexuality (MH) for three reasons: (i) homosexuality in males (HM) is more common than homosexual females; (ii) MH is much more scientifically studied than female homosexuality; and (iii) moral and religious concerns seem much more concentrated on HM than on lesbian behaviour. An impressive amount of empirical data suggests that biology is an important regulator of both heterosexual and homosexual behaviours. Evidence has been produced showing the importance of genetic, autoimmune, and neurohormonal factors in the development of sexual orientation. Criticizing methods and findings produced in the field of biology of sexual orientation 6.

Mustanski et al. admit that genetic research using family and twin methodologies has produced consistent evidence that genes influence sexual orientation, but molecular research has not yet produced compelling evidence for specific genes 7. Although it has been well established that older brothers increase the odds of homosexuality in men, the route by which this occurs has not been fully resolved. Even the robust and elegant evidence solving the Darwinian paradox (how an antireproductive gene may survive?) produced by Camperio-Ciani need to be confirmed in larger samples. This author discusses here the fertility advantages of carrying the "gene" of HM, using arguments similar to that known for the thalassemia trait, which may confer a degree of protection against malaria, prevalent in the regions where the trait is common, thus conferring a selective survival advantage on carriers and perpetuating the mutation

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Male will be included

Exclusion Criteria:

* Patients taking testosterone or its derivative.
* Patients taking anabolic steroids.
* Multi-sexual behaviours.
* HIV patients.
* not having and addictive disorder

Ages: 18 Years to 60 Years | Sex: Male
Age Groups: Adult
Study Population: All individuals with homosexuality from these different locations, Egypt, England, China, and Mexico.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2027-11-20 (Estimated); Study Completion 2028-04-20 (Estimated)

PRIMARY OUTCOMES:
Change of Symptom Checklist-90-Revised (SCL-90-R) from baseline to 34 weeks | from baseline to 34 weeks
  The SCL-90-R Is an inventory developed to assess the intensity of symptoms inventoried during the last weeks. Each of the 90 items that is integrated in the self-report questionnaire is answered in a likert scale from 0 (nothing) to 4 (a lot), depending on the intensity with which the subject has lived in the last weeks the discomfort that each one explores. It is evaluated and interpreted in function of 10 primary dimensions (somatization, obsession-compulsion, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychotic and diverse symptoms and three global indexes of psychological disorders.
Change of Sexual Compulsivity Scale (SCS) from baseline to 34 weeks | from baseline to 34 weeks
  The SCS contains 10 items (e.g., "my desires to have sex have disrupted my daily life"), rated from 1 (not at all like me) to 4 (very much like me). Item responses are summed to derive an overall score (range 10-40). A score of 24 or higher is frequently used to distinguish problematic sexual compulsivity
Change of Safer Sex Self-Efficacy Questionnaire (SSSE) from baseline to 34 weeks | from baseline to 34 weeks
  The 13-item SSSE assesses self-efficacy for condom use in various situations (e.g., "When you really need affection," "When your partner says he/she does not want to use a condom") in response to the prompt, "How confident are you that you could avoid having anal sex without a condom?" using a scale ranging from 1 (not at all tempted) to 5 (extremely tempted). The SSSE predicts condomless anal intercourse among men who have sex with men (MSM; Rendina, 2014).

SECONDARY OUTCOMES:
Change of Measure of Gay-Related Stress (MOGS) from baseline to 34 weeks | from baseline to 34 weeks
  The MOGS contains 56 stressors related to being gay, which participants rated in terms of the negative and positive impact each stressor had if it occurred in the past 12 months along a scale ranging from -3 (extremely negative) to 3 (extremely positive).
Change of Internalized Homophobia Scale (IHP) from baseline to 34 weeks | from baseline to 34 weeks
  The IHP assesses how troubled gay and bisexual men are about their sexual identities over the past year. Participants rate nine items using a scale from 1 (never) to 4 (often). The IHP is associated with general mental and sexual health problems in a sample of adult gay men (Meyer, 1995).
Change of Sexual Orientation Concealment Scale (SOCS) from baseline to 34 weeks | from baseline to 34 weeks
  In the SOCS, participants indicate the degree to which they are "out of the closet" to five domains of people: family; gay, lesbian, and bisexual friends; straight friends; co-workers; and health care providers, using a scale from 1 (out to all) to 4 (out to none).